CLINICAL TRIAL: NCT00844207
Title: A Phase 1, Open Label, Randomized, Single Dose, Parallel Group Study To Estimate The Relative Bioavailability Of Fixed Combination Tablets Of Azithromycin And Chloroquine Compared To Co-Administered Individual Tablets Of Azithromycin And Chloroquine In Healthy Adult Subjects
Brief Title: A Phase 1 Study To Estimate The Relative Bioavailability Of Fixed Combination Tablets Of Azithromycin And Chloroquine Compared To Co-Administered Individual Tablets Of Azithromycin And Chloroquine
Acronym: AZCQ
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: A0661186
Record Dates: First submitted 2009-02-10; First posted 2009-02-16 (Estimated); Last update posted 2009-04-21 (Estimated); Status verified 2009-04

CONDITIONS: Malaria
Keywords: Bioavailability
MeSH Terms: conditions — Malaria | interventions — Chloroquine; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A (Experimental): Two of the fixed combination tablets each containing 250 mg of azithromycin and 155 mg of chloroquine base.
  Interventions: Drug: Fixed combination of Azithromycin and Chloroquine
- Treatment B (Active Comparator): A single tablet containing 500 mg of azithromycin and a single tablet containing 300 mg of chloroquine base.
  Interventions: Drug: Azithromycin and Chloroquine

INTERVENTIONS:
Drug: Fixed combination of Azithromycin and Chloroquine — Pfizer will provide the study medications, fixed combination azithromycin/chloroquine tablets (250 mg/155 mg, base), The study treatment is single dose.
  Arms: Treatment A
Drug: Azithromycin and Chloroquine — Pfizer will provide Zithromax (500 mg) and Aralen (500 mg containing 300 mg chloroquine base). The study treatment is single dose.
  Arms: Treatment B

SUMMARY:
The primary objective is to estimate the relative bioavailability of fixed azithromycin / chloroquine combination tablets relative to co-administered individual tablets of azithromycin and chloroquine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* History of febrile illness within 5 days prior to first dose.
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
AUClast and Cmax of azithromycin and chloroquine for each treatment. | up to 96 hours post dose on Day 5

SECONDARY OUTCOMES:
Tmax of azithromycin and chloroquine for each treatment cohort. | up to 96 hours post dose on Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661186&StudyName=A%20Phase%201%20Study%20To%20Estimate%20The%20Relative%20Bioavailability%20Of%20Fixed%20Combination%20Tablets%20Of%20Azithromycin%20And%20Chloroquine%20Compared%20To%20Co-Adm